CLINICAL TRIAL: NCT02634801
Title: A 24-Week Multicenter, Randomized, Open-Label, Parallel-Group Study Comparing the Efficacy and Safety of Ixekizumab to Fumaric Acid Esters and Methotrexate in Patients With Moderate-to-Severe Plaque Psoriasis Who Are Naive to Systemic Treatment With an Extension Period
Brief Title: A Study of Ixekizumab (LY2439821) in Participants With Moderate-to-Severe Plaque Psoriasis Naive to Systemic Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16190; I1F-EW-RHBZ (Other: Eli Lilly and Company); 2015-002649-69 (EudraCT Number)
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Plaque Psoriasis
Keywords: Fumaderm
MeSH Terms: interventions — Fumarates; Methotrexate; ixekizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: Yes

ARMS (3):
- Ixekizumab (Experimental): 160 milligrams (mg) ixekizumab given as two subcutaneous injections (SC) followed by 80 mg ixekizumab given SC every 2 weeks until week 12 and then 80 mg ixekizumab given SC every 4 weeks until week 24.
  Extension Period: At week 24, participants have the option to continue ixekizumab treatment for up to 36 weeks.
  Interventions: Drug: Ixekizumab
- Fumaric Acid Esters (Active Comparator): Starting dose of 105 mg FAE given orally followed by 215 mg FAE given orally 1 to 3 times per day until week 24.
  Extension Period: At week 24, participants have the option to begin ixekizumab treatment for up to 36 weeks.
  Interventions: Drug: Fumaric Acid Esters; Drug: Ixekizumab
- Methotrexate (Active Comparator): 7.5 mg starting dose up to 30 mg MTX given orally once a week until week 24.
  Extension Period: At week 24, participants have the option to begin ixekizumab treatment for up to 36 weeks.
  Interventions: Drug: Methotrexate; Drug: Ixekizumab

INTERVENTIONS:
Drug: Fumaric Acid Esters — Administered orally
  Arms: Fumaric Acid Esters
Drug: Methotrexate — Administered orally
  Arms: Methotrexate
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821

SUMMARY:
The main purpose of this study is to evaluate the efficacy of ixekizumab compared to fumaric acid esters (FAE) and methotrexate (MTX) in participants with moderate-to-severe plaque psoriasis who are naive to systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Present with moderate-to-severe chronic plaque psoriasis based on a diagnosis of chronic psoriasis for at least 6 months before baseline.
* Participants who are candidates for systemic therapy and who are naive to systemic treatment for psoriasis.
* Have a (PASI score >10 or BSA >10) and DLQI >10 at screening and at baseline.

Exclusion Criteria:

* Have predominant pattern of pustular, erythrodermic, and/or guttate forms of psoriasis.
* Have received systemic nonbiologic psoriasis therapy.
* Have prior, concurrent, or recent use of ixekizumab or any other biological psoriasis therapy.
* Have any condition or contraindication as addressed in the local labeling for MTX or FAE.
* Presence of significant uncontrolled cerebro-cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, neurologic, or neuropsychiatric disorders or abnormal laboratory values at screening.
* Have severe gastrointestinal disease, oral ulcer, or known, active gastrointestinal ulcer.
* Have had a serious infection or are immunocompromised.
* At screening, participants with significant, present, or early liver disease, e.g., explained by alcohol consumption or hepatic insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2016-11-29 (Actual); Study Completion 2017-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (21):
- Germany (21):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augsburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bochum
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bonn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buxtehude
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erlangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Friedrichshafen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gelsenkirchen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanau
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Kiel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lübeck
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Selters
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stuttgart
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tübingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Reich K, Augustin M, Thaci D, Pinter A, Leutz A, Henneges C, Schneider E, Schacht A, Dossenbach M, Mrowietz U. A 24-week multicentre, randomized, open-label, parallel-group study comparing the efficacy and safety of ixekizumab vs. fumaric acid esters and methotrexate in patients with moderate-to-severe plaque psoriasis naive to systemic treatment. Br J Dermatol. 2020 Apr;182(4):869-879. doi: 10.1111/bjd.18384. Epub 2019 Nov 19. PMID 31376153

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment Period (Weeks 0 to 24), Extension Period (Weeks 24 to 36) followed by post-treatment follow-up period occurring from last treatment visit (week 36), or Early Termination Visit (ETV) up to a minimum of 12 weeks following that visit.
Groups:
- Fumaric Acid Esters: Starting dose of 105 mg Fumaric Acid Esters (FAE) given orally followed by 215 mg FAE given orally 1 to 3 times per day until week 24.
  Extension Period: At week 24, participants have the option to begin ixekizumab treatment for up to 36 weeks.
- Methotrexate: 7.5 mg starting dose up to 30 mg Methotrexate (MTX) given orally once a week until week 24.
  Extension Period: At week 24, participants have the option to begin ixekizumab treatment for up to 36 weeks.
Period: Treatment Period (Weeks 0 to 24)
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Started | 54 | 54 | 54
Received at Least 1 Dose of Study Drug | 54 | 52 | 52
Completed | 50 | 23 | 49
Not Completed | 4 | 31 | 5
Not completed — Adverse Event | 2 | 20 | 0
Not completed — Lack of Efficacy | 0 | 2 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 8 | 3
Period: Extension Period (Weeks 24 to 36)
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Started | 48 (Participants had the option to enter the Extension Period or proceed directly to the Followup Period) | 19 (Participants had the option to enter the Extension Period or proceed directly to the Followup Period) | 31 (Participants had the option to enter the Extension Period or proceed directly to the Followup Period)
Completed | 45 | 18 | 29
Not Completed | 3 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Missing | 1 | 0 | 0
Period: Follow-up Period
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Started | 41 (Participants who discontinued previous periods had option to enter post treatment follow-up period.) | 26 (Participants who discontinued previous periods had option to enter post treatment follow-up period.) | 46 (Participants who discontinued previous periods had option to enter post treatment follow-up period.)
Completed | 36 | 18 | 38
Not Completed | 5 | 8 | 8
Not completed — Lost to Follow-up | 3 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 5
Not completed — Adverse Event | 1 | 5 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who had baseline data.
Groups:
- Ixekizumab: 160 mg ixekizumab given as two SC injection followed by 80 mg ixekizumab given SC every 2 weeks until week 12 and then 80 mg ixekizumab given SC every 4 weeks until week 24.
  Extension Period: At week 24, participants have the option to continue ixekizumab treatment for up to 36 weeks.
- Total: Total of all reporting groups
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate | Total
Number analyzed (Participants) | 54 | 54 | 54 | 162
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All randomized participants who had baseline data.
  Years
    number analyzed (Participants) | 54 | 52 | 52 | 158
    (all) | 44.3 (13.84) | 43.1 (14.16) | 38.7 (12.90) | 42.1 (13.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 18 | 41
  Male | 42 | 43 | 36 | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 43 | 44 | 42 | 129
  More than one race | 10 | 10 | 9 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 54 | 54 | 54 | 162

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥75% Improvement in Psoriasis Area and Severity Index (PASI 75) at Week 24
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored separately and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs (0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease).
Time Frame: Week 24
Population: All randomized participants who had a post-baseline measurement for PASI 75. Participants who did not meet the clinical response criteria or had missing data were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number; unit: Percentage of Participants
Groups:
- Ixekizumab: 160 mg ixekizumab given as two SC injections followed by 80 mg ixekizumab given SC every 2 weeks until week 12 and then 80 mg ixekizumab given SC every 4 weeks until week 24.
  Extension Period: At week 24, participants have the option to continue ixekizumab treatment for up to 36 weeks.
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 54 | 54 | 54
Percentage of Participants | 90.7 | 22.2 | 70.4
Statistical Analysis 1: Comparison: Ixekizumab vs Fumaric Acid Esters; Test type: Superiority or Other; p < .0001, Fisher Exact; Risk Ratio (RR) = 4.08, 95% CI 2-sided [2.46 to 6.77]
Statistical Analysis 2: Comparison: Ixekizumab vs Methotrexate; Test type: Superiority or Other; p = 0.0137, Fisher Exact; Risk Ratio (RR) = 1.29, 95% CI 2-sided [1.06 to 1.56]

2. Secondary Outcome: Percentage of Participants With a ≥90% Improvement in Psoriasis Area and Severity Index (PASI 90) From Baseline
Description: as for outcome 1
Time Frame: Week 24
Population: All randomized participants who had a post-baseline measurement for PASI 90. Participants who did not meet the clinical response criteria or had missing data were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 54 | 54 | 54
Percentage of Participants | 79.6 | 9.3 | 38.9

3. Secondary Outcome: Percentage of Participants With a 100% Improvement in Psoriasis Area and Severity Index (PASI 100) From Baseline
Description: as for outcome 1
Time Frame: Week 24
Population: All randomized participants who had a post-baseline measurement for PASI 100. Participants who did not meet the clinical response criteria or had missing data were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 54 | 54 | 54
Percentage of Participants | 40.7 | 3.7 | 13.0

4. Secondary Outcome: Change From Baseline in PASI Total Score
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored separately and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs (0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease). LS mean change from baseline in PASI was calculated using Analysis of Covariance (ANCOVA) with modified Baseline- Observation- Carried Forward (mBOCF) and with terms for baseline and treatment.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for PASI.
  mBOCF: Participants who discontinued treatment due to Adverse Event (AE) were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 54 | 50 | 52
units on a scale | -16.68 [-18.46 to -14.91] | -4.93 [-6.78 to -3.09] | -14.61 [-16.42 to -12.80]

5. Secondary Outcome: Percentage of Participants With a Static Physician Global Assessment (sPGA) (0,1) and ≥2 Point Improvement From Baseline Among Those With sPGA Score ≥3 at Baseline
Description: The sPGA is the physician's determination of the participant's Psoriasis (Ps) lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participants Ps were assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe). An sPGA responder was defined as having a post-baseline sPGA score of "0" or "1" with at least a 2-point improvement from baseline.
Time Frame: Week 24
Population: All randomized participants with baseline sPGA >=3 & received at least 1 dose of study drug and had a post-baseline measurement for sPGA. Participants who did not meet the clinical response criteria or had missing data were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 52 | 53 | 52
Percentage of Participants | 86.5 | 13.2 | 51.9

6. Secondary Outcome: Percentage of Participants Achieving DLQI (0,1)
Description: The DLQI is a simple, participant-administered, 10 question, validated, quality-of-life questionnaire that covers 6 domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include "not at all," "a lot," and "very much," with corresponding scores of 1, 2, and 3, respectively, and unanswered ("not relevant") responses scored as "0." Totals range from 0 to 30 (less to more impairment), and a 5-point change from baseline is considered clinically relevant.
Time Frame: Week 24
Population: All randomized participants who had a post-baseline measurement for DLQI. Participants who did not meet the clinical response criteria or had missing data were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 54 | 54 | 54
Percentage of Participants | 63.0 | 14.8 | 37.0

7. Secondary Outcome: Change From Baseline on Dermatology Life Quality Index (DLQI) Total Score
Description: The DLQI is a simple, participant-administered, 10 question, validated, quality-of-life questionnaire that covers 6 domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include "not at all," "a lot," and "very much," with corresponding scores of 1, 2, and 3, respectively, and unanswered ("not relevant") responses scored as "0." Totals range from 0 to 30 (less to more impairment), and a 5-point change from baseline is considered clinically relevant. LS mean change from baseline in DLQI was calculated using ANCOVA with mBOCF and with terms for baseline and treatment.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for DLQI.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 52 | 49 | 49
units on a scale | -13.08 [-14.56 to -11.61] | -5.37 [-6.88 to -3.86] | -12.81 [-14.32 to -11.29]

8. Secondary Outcome: Change From Baseline in Body Surface Area (BSA) Affected by Psoriasis
Description: The percentage involvement of psoriasis on each participant's body surface area was assessed by the investigator on a continuous scale from 0% (no involvement) to 100% (full involvement), in which 1% corresponds to the size of the participant's hand including palm, fingers and thumb.
  LS mean change from baseline in BSA was calculated using ANCOVA with mBOCF and with terms for baseline and treatment.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for BSA.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: % Body Surface Affected
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 54 | 50 | 52
% Body Surface Affected | -20.64 [-23.21 to -18.08] | -5.26 [-7.93 to -2.60] | -18.46 [-21.08 to -15.85]

9. Secondary Outcome: Change From Baseline in Palmoplantar Psoriasis Severity Index (PPASI) Total Score
Description: The Palmoplantar PASI is a composite score derived from the sum scores for erythema, induration, and desquamation multiplied by a score for the extent of palm and sole area involvement, ranging from 0 (no PPASI) to 72 (most severe PPASI). The PPASI was only assessed if participants have palmoplantar psoriasis at baseline.
  LS mean change from baseline in PPASI was calculated using ANCOVA with mBOCF and with terms for baseline and treatment.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for PPASI.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 12 | 14 | 9
units on a scale | -7.23 [-10.88 to -3.59] | -2.45 [-6.03 to 1.13] | -3.77 [-8.10 to 0.56]

10. Secondary Outcome: Change From Baseline in Psoriasis Scalp Severity Index (PSSI) Total Score
Description: The PSSI is a physician assessment of erythema, induration and desquamation and percent of scalp that is covered with a scores range from 0 (none) to 4 (very severe). The composite score is derived from the sum of scores for erythema, induration, and desquamation multiplied by the score recorded for the extent of the scalp area involved, 1 (<10%) to 6 (90%-100%) with a total score ranging from 0 (less severity) to 72 (more severity).
  LS mean change from baseline in PSSI was calculated using ANCOVA with mBOCF and with terms for baseline and treatment.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for Psoriasis Scalp.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 40 | 39 | 40
units on a scale | -20.85 [-23.63 to -18.06] | -6.76 [-9.58 to -3.94] | -18.56 [-21.35 to -15.78]

11. Secondary Outcome: Patient Benefit Index (PBI) Overall Benefit Score
Description: The PBI assessment consists of 2 steps: before treatment, every patient defines his/her treatment needs according to a standardized list (Patient Needs Questionnaire [PNQ]). After treatment, the patient rates the degree of benefits achieved (Patient Benefits Questionnaire [PBQ]). 25 items are rated on a 5-point scale with values from 0 (not at all) to 4 (very), allowing for "did not apply to me" (5) and missing.
  For each treatment goal the PNQ importance is derived by dividing the respective PNQ item by the sum of all PNQ items. The weighted sum of each PBQ item with its respective PNQ importance yields the PBI score.
  LS mean was calculated using ANCOVA with LOCF and with a term for treatment.
Time Frame: Week 24
Population: All randomized participants who received at least 1 dose of study drug and had a baseline PBI questionnaire such that postbaseline PBI assessments can be valid (nonmissing).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 43 | 41 | 50
units on a scale | 3.42 [2.99 to 3.84] | 2.33 [1.81 to 2.84] | 2.66 [2.23 to 3.10]

12. Secondary Outcome: Change From Baseline on Itch Numeric Rating Scale (NRS) Score
Description: The Itch NRS is a participant-administered single-item 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching from psoriasis (Ps) is indicated by circling the number that best describes the worst level of itching in the past 24 hours.
  LS mean change from baseline was calculated using ANCOVA with mBOCF and with terms for baseline and treatment.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for Itch NRS score.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 53 | 50 | 52
units on a scale | -5.25 [-5.89 to -4.61] | -1.50 [-2.15 to -0.84] | -4.40 [-5.05 to -3.76]

13. Secondary Outcome: Change From Baseline on the Skin Pain Visual Analog Scale (VAS)
Description: The pain VAS is a participant-administered single-item scale designed to measure Skin pain from Psoriasis using a 100 millimeter (mm) horizontal VAS. Overall severity of participant's skin pain from Psoriasis is indicated by placing a single mark on the horizontal 100 mm scale from 0 mm (no pain) to 100 mm (pain as severe as you can imagine).
  LS mean change from baseline was calculated using ANCOVA with mBOCF and with terms for baseline and treatment.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for skin pain VAS.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Millimeter (mm)
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 53 | 50 | 52
Millimeter (mm) | -33.83 [-39.46 to -28.20] | -7.20 [-12.99 to -1.42] | -28.29 [-33.98 to -22.60]

14. Secondary Outcome: Change From Baseline on Quick Inventory of Depressive Symptomatology-Self Report (16 Items) (QIDS-SR16)
Description: QIDS-SR16 is a participant-administered, 16-item instrument intended to assess the existence and severity of symptoms of depression. A participant is asked to consider each statement as it relates to the way they have felt for the past 7 days and rate each on a 4-point scale: 0 (best) to 3 (worst). The sum of the 16 items corresponding to 9 depression domains [sad mood, concentration, self-criticism, suicidal ideation, interest, energy/fatigue, sleep disturbance (initial, middle and late insomnia or hypersomnia), decrease/increase in appetite/weight, and psychomotor agitation/retardation] to give a single total scores range from 0 to 27, with higher scores indicating greater symptom severity. Whereas 0-5 indicates no symptoms.
  LS mean change from baseline was calculated using ANCOVA with mBOCF and with terms for baseline and treatment.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for QIDS-SR16.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 51 | 49 | 50
units on a scale | -2.16 [-3.00 to -1.32] | -1.01 [-1.89 to -0.14] | -2.50 [-3.37 to -1.64]

15. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS)
Description: The SF-36 is a participant-reported outcome measure evaluating participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. The 8 domains are regrouped into the PCS and MCS scores. The summary scores range from 0 to 100, lower scores = more disability, higher scores = less disability and better health. In this study, the SF-36 acute version was used, which has a 1-week recall period.
  LS mean change from baseline was calculated using ANCOVA with mBOCF and with terms for baseline and treatment.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for SF36 PCS score.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 50 | 48 | 49
units on a scale | 4.45 [2.29 to 6.60] | 0.57 [-1.64 to 2.77] | 4.01 [1.83 to 6.19]

16. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Mental Component Summary (MCS) Scores
Description: as for outcome 15
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for SF36 MCS score.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 50 | 48 | 49
units on a scale | 7.13 [4.99 to 9.27] | 3.39 [1.19 to 5.59] | 6.99 [4.80 to 9.17]

17. Secondary Outcome: Change From Baseline on Patient's Global Assessment (PatGA) of Disease Severity
Description: The PatGA is a single-item self-reported instrument asking the participant to rate the severity of their psoriasis "today" by circling a number on the numeric rating scale from 0 (Clear = no psoriasis) to 5 (Severe = the worst their psoriasis has ever been).
  LS mean change from baseline was calculated using ANCOVA with mBOCF and with terms for baseline and treatment.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for PatGA.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 54 | 50 | 50
units on a scale | -3.12 [-3.47 to -2.78] | -0.87 [-1.23 to -0.51] | -2.39 [-2.75 to -2.04]

18. Secondary Outcome: Change From Baseline on the Psoriasis Skin Appearance Bothersomeness (PSAB) Total Score
Description: PSAB measure is a 3-item scale designed to measure the degree of bothersomeness of skin appearance due to Ps in participants with Ps. Participants are asked to indicate on 3 numeric rating scales (NRS) from 0 (not at all bothered) to 10 (extremely bothered) how bothered they are by any redness or discoloration, thickness, and scaling or flaking on their skin due to Ps.
  The scores from the 3 NRS items are summed for a total score ranging from 0 to 30, where 0 indicating no bothersomeness and 30 indicating greater bothersomeness.
  LS mean change from baseline was calculated using ANCOVA with mBOCF and with terms for baseline and treatment.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for PSAB.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 52 | 47 | 48
units on a scale | -19.87 [-22.38 to 17.36] | -5.18 [-7.82 to -2.54] | -15.05 [-17.67 to -12.43]

19. Secondary Outcome: Change From Baseline on the Nail Assessment in Psoriasis and Psoriatic Arthritis (NAPPA-CLIN) Total Score
Description: NAPPA is a clinical and participant-reported outcomes tool, and consists of 3 components: a questionnaire assessing nail-specific quality of life NAPPA-QoL (Nail Assessment in Psoriasis and Psoriatic Arthritis Quality of Life), a 2-part questionnaire assessing participant relevant needs and treatment benefits NAPPA-PBI (Nail Assessment in Psoriasis and Psoriatic Arthritis - Patient Benefit Index), and a clinical assessment of objective finger nail psoriasis severity NAPPA-CLIN.
  Sum of all assessed finger and toes ranging between 0 (no involvement) to 16 (worst involvement).
  LS mean change from baseline was calculated using ANCOVA with mBOCF and with terms for baseline and treatment.
Time Frame: Baseline, Week 24
Population: All randomized participants who had palmoplantar, scalp, or nail involvement at baseline.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 35 | 29 | 27
units on a scale | -6.58 [-8.12 to -5.04] | -0.14 [-1.91 to 1.62] | -3.41 [-5.30 to -1.52]

20. Secondary Outcome: Change From Baseline in European Quality of Life - 5 Dimensions 5 Level (EQ-5D) + Bolt On UK Population-based Index Score
Description: The European Quality of Life - 5 Dimensions 5 Level (EQ-5D-5L) is a standardized measure of health status used to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D-5L consists of a descriptive system of the respondent's health which comprises the following 5 dimensions: 1) mobility 2) self-care 3) usual activities 4) pain/discomfort 5) anxiety/depression. The EQ-5D-5L health states were converted into a single summary index by applying a crosswalk using a United Kingdom (UK) Population value set to each of the levels in each dimension. This produced participant-level index scores between -0.594 and 1.0 (worse to better health).
  LS mean change from baseline was calculated using ANCOVA with mBOCF and with terms for baseline and treatment.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for EQ-5D 5L Index.mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 52 | 47 | 50
units on a scale | 0.15 [0.11 to 0.20] | 0.04 [-0.01 to 0.09] | 0.15 [0.10 to 0.20]

21. Secondary Outcome: Change From Baseline in European Quality of Life - 5 Dimensions 5 Level (EQ-5D 5L) "Bolt On" - Psoriasis (PSO) Index Score
Description: The European Quality of Life - 5 Dimensions 5 Level (EQ-5D-5L) is a standardized measure of health status used to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D-5L consists of a descriptive system of the respondent's health which comprises the following 5 dimensions: 1) mobility 2) self-care 3) usual activities 4) pain/discomfort 5) anxiety/depression. The Bolt On PSO is an addition to the EQ-5D-5L that consists of 2 dimensions specific to psoriatic disease: 6) skin irritation (itching) and 7) self-confidence. Index scores for the Bolt On PSO range from 0.0042 to 1.0 (worse to better health).
  LS mean change from baseline was calculated using ANCOVA with mBOCF and with terms for baseline and treatment.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for EQ-5D 5L "Bolt On" PSO-Index.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 52 | 46 | 50
units on a scale | 0.15 [0.12 to 0.18] | 0.05 [0.01 to 0.08] | 0.13 [0.10 to 0.16]

22. Secondary Outcome: Change From Baseline in European Quality of Life - 5 Dimensions 5 Level (EQ-5D 5L) "Bolt On" - Visual Analog Scale Score
Description: The EQ-5D 5L is a standardized measure of health status that includes a descriptive system of the respondent's health and a rating of his/her current health state using a 0 (worst health imaginable)- to 100 (best health imaginable)-millimeter (mm) Visual Analog Scale (VAS).
  LS mean change from baseline was calculated using ANCOVA with mBOCF and with terms for baseline and treatment.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for EQ-5D 5L + Bolt on VAS.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Millimeter (mm)
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 52 | 48 | 50
Millimeter (mm) | 16.91 [12.23 to 21.59] | 6.08 [1.21 to 10.96] | 13.91 [9.14 to 18.69]

23. Secondary Outcome: Change From Baseline on the Work Productivity Activity Impairment Questionnaire-Psoriasis (WPAI-PSO), Absenteeism Score
Description: The WPAI-PSO consists of 6 questions to determine employment status, hours missed from work because of psoriasis, hours missed from work for other reasons, hours actually worked, the degree to which psoriasis affected work productivity while at work, and the degree to which psoriasis affected activities outside of work. Four scores are derived: percentage of absenteeism, percentage of presenteeism (reduced productivity while at work), an overall work impairment score that combines absenteeism and presenteeism, and percentage of impairment in activities performed outside of work. Each WPAI score is expressed as impairment percentages (0-100), where 0 (no impairement) and 100 (greater impairment).
  LS mean change from baseline was calculated using ANCOVA with mBOCF and with terms for baseline and treatment.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for WPAI-PSO absenteeism score.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 26 | 30 | 39
units on a scale | 3.08 [-3.79 to 9.96] | -1.26 [-7.69 to 5.17] | 0.06 [-5.49 to 5.62]

24. Secondary Outcome: Change From Baseline on the Work Productivity Activity Impairment Questionnaire-Psoriasis (WPAI-PSO), Presenteeism Score
Description: as for outcome 23
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for WPAI-PSO Presenteeism score.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 29 | 32 | 39
units on a scale | -22.70 [-28.73 to -16.66] | -5.29 [-11.10 to 0.52] | -20.32 [-25.51 to -15.13]

25. Secondary Outcome: Change From Baseline on the Work Productivity Activity Impairment Questionnaire-Psoriasis (WPAI-PSO), Impairment in Activities Performed Outside of Work
Description: as for outcome 23
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for WPAI-PSO.
  mBOCF: Participants who discontinued treatment due to AE were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 53 | 50 | 48
units on a scale | -28.23 [-33.99 to -22.47] | -3.45 [-9.38 to 2.47] | -23.57 [-29.58 to -17.55]

26. Secondary Outcome: Change From Baseline on the Work Productivity Activity Impairment Questionnaire-Psoriasis (WPAI-PSO), Overall Work Impairment Score
Description: as for outcome 23
Time Frame: Baseline, Week 24
Population: as for outcome 25
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 25 | 30 | 38
units on a scale | -18.20 [-26.29 to -10.11] | -6.20 [-13.66 to 1.27] | -19.80 [-26.31 to -13.29]

27. Secondary Outcome: Percentage of Participants With Positive Responses to Neck/Face Psoriasis Question
Description: Studying psoriasis involvement in the face, neck, and the genitals is of considerable interest for participants. These are locations that bear high potential for stigmatization and/or psychological distress, and, hence, effects in those regions are assumed to heavily influence participant's quality of life.
  Following set of binary questions were asked to check the satisfaction of participants.
  1. Does the participant currently have visible psoriasis on face/neck? (Yes/No)
  2. Does the participant currently have psoriasis on the genital area? (Yes/No)
Time Frame: Week 24
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for binary questions.
  Participants who did not meet the clinical response criteria or had missing data were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 33 | 34 | 36
Percentage of Participants | 81.8 | 26.5 | 66.7

28. Secondary Outcome: Percentage of Participants Positive Responses to Genital Psoriasis Question
Description: Studying psoriasis involvement in the face, neck, and the genitals is of considerable interest for participants. These are locations that bear high potential for stigmatization and/or psychological distress, and, hence, effects in those regions are assumed to heavily influence participant's quality of life.
  Following set of binary questions were asked to check the satisfaction of participants.
  1. Does the patient currently have visible psoriasis on face/neck? (Yes/No)
  2. Does the patient currently have psoriasis on the genital area? (Yes/No) The genital area includes the labia majora (hair-bearing), labia minora modified mucus membrane, and perineum in female patients; and the penis glans, penis - shaft, and scrotum in male patients.
Time Frame: Week 24
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 20 | 24 | 24
Percentage of participants | 85.0 | 29.2 | 75.0

29. Secondary Outcome: Mean Adherence on Medication and Satisfaction With Therapy (STAQ)
Description: Systemic Therapy Adherence Questionnaire (STAQ) is a 38 item questionnaire that was developed by shortening and adapting the Topical Treatment Adherence Questionnaire (TTAQ) for administration to participants under systemic therapy. The following STAQ items are of special interest for this study.
  1. STAQ item 13 (The treatment does not affect my sex life)
  2. STAQ item 16 (I am enjoying life again as a result of the treatment)
  3. STAQ item 20 (The side effects of the treatment were acceptable)
  4. STAQ item 31 (I am satisfied with the efficacy of the treatment)
  5. STAQ item 32 (I am satisfied with the tolerability of the treatment)
  6. STAQ item 35 (The positive aspects of the treatment outweigh the negative ones).
  The STAQ items are on a 4-point Likert scale with scores between 0 (strong disagreement) and 3 (strong agreement). LS mean was calculated using ANCOVA with term for treatment.
Time Frame: Week 24
Population: All randomized participants who received at least 1 dose of study drug and had a post-baseline measurement for Systemic Therapy Adherence Questionnaire (STAQ).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixekizumab | Fumaric Acid Esters | Methotrexate
Number analyzed (Participants) | 49 | 22 | 48
units on a scale
  STAQ item 13: number analyzed (Participants) | 44 | 20 | 40
  STAQ item 13 | 2.84 [2.68 to 3.00] | 2.75 [2.51 to 2.99] | 2.78 [2.61 to 2.94]
  STAQ item 16: number analyzed (Participants) | 45 | 21 | 42
  STAQ item 16 | 2.82 [2.60 to 3.04] | 2.00 [1.68 to 2.32] | 2.43 [2.20 to 2.66]
  STAQ item 20: number analyzed (Participants) | 42 | 22 | 43
  STAQ item 20 | 2.76 [2.51 to 3.01] | 2.00 [1.66 to 2.34] | 2.42 [2.17 to 2.66]
  STAQ item 31 | 2.88 [2.68 to 3.08] | 2.09 [1.79 to 2.39] | 2.29 [2.09 to 2.50]
  STAQ item 32 | 2.86 [2.66 to 3.05] | 1.95 [1.66 to 2.25] | 2.50 [2.30 to 2.70]
  STAQ item 35: number analyzed (Participants) | 45 | 22 | 47
  STAQ item 35 | 2.80 [2.58 to 3.02] | 2.14 [1.82 to 2.46] | 2.53 [2.31 to 2.75]

ADVERSE EVENTS:
Time Frame: Up to 48 Weeks
Description: All the randomized participants who received at least one dose of the study drug.
Groups:
- Ixekizumab-Treatment Period; Ixekizumab-Extension Period: 160 milligrams (mg) ixekizumab given as two subcutaneous injections (SC) followed by 80 mg ixekizumab given SC every 2 weeks until week 12 and then 80 mg ixekizumab given SC every 4 weeks until week 24.
  Extension Period: At week 24, participants have the option to continue ixekizumab treatment for up to 36 weeks.
- Fumaric Acid Esters-Treatment Period; Fumaric Acid Esters-Extension Period: Starting dose of 105 mg FAE given orally followed by 215 mg FAE given orally 1 to 3 times per day until week 24.
  Extension Period: At week 24, participants have the option to begin ixekizumab treatment for up to 36 weeks.
- Methotrexate-Treatment Period; Methotrexate-Extension Period: 7.5 mg starting dose up to 30 mg MTX given orally once a week until week 24. Extension Period: At week 24, participants have the option to begin ixekizumab treatment for up to 36 weeks.
- Follow-up Period: Participants were allowed to continue the treatment administered during the treatment and extension period.
Arm/Group | Ixekizumab-Treatment Period | Fumaric Acid Esters-Treatment Period | Methotrexate-Treatment Period | Ixekizumab-Extension Period | Fumaric Acid Esters-Extension Period | Methotrexate-Extension Period | Follow-up Period
Serious Adverse Events (participants affected / at risk) | 1/54 | 3/52 | 1/52 | 3/48 | 1/19 | 4/31 | 4/113
Other Adverse Events (participants affected / at risk) | 37/54 | 39/52 | 38/52 | 24/48 | 15/19 | 18/31 | 0/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixekizumab-Treatment Period (N=54) | Fumaric Acid Esters-Treatment Period (N=52) | Methotrexate-Treatment Period (N=52) | Ixekizumab-Extension Period (N=48) | Fumaric Acid Esters-Extension Period (N=19) | Methotrexate-Extension Period (N=31) | Follow-up Period (N=113)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixekizumab-Treatment Period (N=54) | Fumaric Acid Esters-Treatment Period (N=52) | Methotrexate-Treatment Period (N=52) | Ixekizumab-Extension Period (N=48) | Fumaric Acid Esters-Extension Period (N=19) | Methotrexate-Extension Period (N=31) | Follow-up Period (N=113)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 3 (3) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 19 (26) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 24 (29) | 6 (6) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 5 (14) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral mucosal eruption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 3 (3) | 8 (14) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (10) | 3 (13) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 7 (23) | 0 (0) | 0 (0) | 1 (9) | 3 (6) | 6 (31) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (10) | 3 (9) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 20 (23) | 9 (13) | 18 (21) | 18 (25) | 6 (7) | 10 (15) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 4 (6) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 7 (7) | 4 (4) | 9 (12) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (2) | 2 (2) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Xanthelasma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 13 (19) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days